CLINICAL TRIAL: NCT06150469
Title: Efficacy of Ginger and Lemon Essential Oil Inhalation on Chemotherapy-induced Nausea and Vomiting in Patients with Haematological Malignancies: a Multicenter, Double-blind, Randomised Controlled Trial
Brief Title: Efficacy of Inhaled Aromatherapy on Nausea and Vomiting in Hematological Malignancies
Acronym: AROM-HEMATO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 87RI23_0013-AROM-HEMATO
Record Dates: First submitted 2023-09-07; First posted 2023-11-29 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Double-blind randomised controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blend of ginger and lemon essential oils (Active Comparator): The experimental group will benefit from conventional management of NVCI (antiemetic prophylaxis in accordance with ESMO international recommendations) plus an aromastick of ginger and lemon essential oils renewed with each course of chemotherapy.
  Patients were included for 3 cycles of chemotherapy (C1, C2, C3).
  Interventions: Combination Product: "Blend of ginger and lemon essential oils", "Neutral oil"
- Neutral oil (Placebo Comparator): The control group will receive conventional management (antiemetic prophylaxis according to international recommendations, ESMO) of NVCI plus a placebo of aromastick containing a neutral, odourless oil, renewed with each course of chemotherapy.
  Interventions: Combination Product: "Blend of ginger and lemon essential oils", "Neutral oil"

INTERVENTIONS:
Combination Product: "Blend of ginger and lemon essential oils", "Neutral oil" — Patients will be given aromasticks to inhale the blend of essential oils.

SUMMARY:
This project will optimise the management of chemotherapy-induced nausea and vomiting, with improvements in nausea and vomiting scores, quality of life and appetite expected in participants benefiting from the intervention. In all cases, the use of complementary methods is recommended and improves the management of people with cancer because they offer a person-centred approach.

DETAILED DESCRIPTION:
The aim is to evaluate the efficacy of inhalation of a mixture of ginger and lemon Essential Oils (EO) versus placebo in addition to conventional antiemetic treatments on the intensity of chemo-induced nausea during the acute phase D1 (H24) of its onset in patients with C1 haematological malignancies.

This multicentre study will be carried out in 5 establishments (haematology and oncology care sectors), which represents a very high potential for inclusion.

In addition, the investigator expect a very high acceptance rate for this study. In fact, in the context of CINV, this care strategy may meet a patient's expectation of symptoms (nausea, vomiting) that they find difficult to manage. Finally, it is known that patients in these care sectors are very keen on supportive care to improve their quality of life, so this is a potentially very interesting opportunity without any particular risk that is offered to participants in this study.

A nurse and a doctor with a postgraduate diploma in aromatherapy are coordinating the team, with the support of a nurse trained in evidence-based practice research methodology. Institutional procedures drawn up by the team at Limoges University Hospital describe the general procedure for using aromatherapy in a scientific and safe way, the protocols that can be used to describe the operating methods, the traceability of the manufacture of the mixtures and their administration, and the evaluation of their effectiveness. Supporting documents, an information note and a monitoring sheet have been created and are being used.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years,
* Chemo-naive patients at inclusion,
* Patients with haematological malignancies treated treated with chemotherapy,
* Patients physically and mentally able to use the aromastick,
* Patients who speak, read and write French,
* Patients who have given signed consent,
* Patients with social security cover.

Exclusion Criteria:

* Asthmatic patients.
* Patients with anosmia.
* Patients allergic to EO, lemon or ginger.
* Patients who have already received aromatherapy to treat chemotherapy-induced nausea and vomiting,
* Patients practising herbal medicine or acupuncture,
* Pregnant and breast-feeding women,
* Patients under guardianship, tutorship or curatorship,
* Patients taking part in interventional studies involving antiemetic drugs or nutritional products,
* Patients who have already had cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-12-16 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Efficacy of inhaled aromatherapy on acute nausea | 1 month, 2 months and 3 months
  To assess difference of nausea intensity score measured by MAT Tool between groups oils (EO) of ginger and lemon versus placebo in addition to addition to conventional antiemetic treatments on intensity of chemo-induced nausea during the acute phase D1 (H24) of onset in patients with haematological malignancies C1 haematological malignancies.
  MAT is used to self-assess the prevention and control of chemotherapy-induced nausea and vomiting. It comprises 2 evaluation parts: the first is a Likert scale assessing the intensity of chemotherapy-induced nausea (0-10), and the second is a record of the frequency of vomiting in the acute (H24) and delayed (H96) phases of chemo-induced nausea and vomiting onset.

SECONDARY OUTCOMES:
Efficacy of inhaled aromatherapy on vomiting frequency | 1 day, 1 month
  To evaluate difference of vomiting fréquency measure by MAT Tool between groups.
  MAT is used to self-assess the prevention and control of chemotherapy-induced nausea and vomiting. It comprises 2 evaluation parts: the first is a Likert scale assessing the intensity of chemotherapy-induced nausea (0-10), and the second is a record of the frequency of vomiting in the acute (H24) and delayed (H96) phases of chemo-induced nausea and vomiting onset.
Efficacy of inhaled aromatherapy on acute nausea between 4 days and 1 month | 4 days, 1 month
  To assess difference of nausea intensity score measured by MAT Tool between groups.
  MAT is used to self-assess the prevention and control of chemotherapy-induced nausea and vomiting. It comprises 2 evaluation parts: the first is a Likert scale assessing the intensity of chemotherapy-induced nausea (0-10), and the second is a record of the frequency of vomiting in the acute (H24) and delayed (H96) phases of chemo-induced nausea and vomiting onset.
Efficacy of inhaled aromatherapy on vomiting frequency between 4 days and 1 month | 4 days, 1 month
  To evaluate difference of vomiting fréquency measure by MAT Tool between groups.
  MAT is used to self-assess the prevention and control of chemotherapy-induced nausea and vomiting. It comprises 2 evaluation parts: the first is a Likert scale assessing the intensity of chemotherapy-induced nausea (0-10), and the second is a record of the frequency of vomiting in the acute (H24) and delayed (H96) phases of chemo-induced nausea and vomiting onset.
Efficacy of inhaled aromatherapy | 1 month, 2 months and 3 months
  To compare the efficacy of inhaled aromatherapy on the evolution of nausea intensity in the acute phase acute phase (D1) and then the delayed phase (D4) chemotherapy cycles (C1, C2 and C3).
  MAT is used to self-assess the prevention and control of chemotherapy-induced nausea and vomiting. It comprises 2 evaluation parts: the first is a Likert scale assessing the intensity of chemotherapy-induced nausea (0-10), and the second is a record of the frequency of vomiting in the acute (H24) and delayed (H96) phases of chemo-induced nausea and vomiting onset.
Anticipatory nausea | 1 month, 2 months and 3 months
  Compare the intensity of chemo-induced nausea. Compared the mean difference of anticipatory nausea intensity score measured by a Likert scale (ranging from 0-10 with zéro none and 10 as much as possible) between groups before the start of each cycle of chemotherapy (C1, C2, C3) between groups.
Compare the proportion of chemically-induced emesis | 1 month, 2 months and 3 months
  Compare the proportion of chemically-induced emesis before the start of each cycle of chemotherapy (C1, C2, C3) between groups.
Independent determinants of the presence of nausea then vomiting | 1 month, 2 months and 3 months
  To identify, in patients who received aromatherapy, the association between independent determinants of the presence of nausea then vomiting at the acute phase (D1) and at the delayed phase (D4) of the first cycle of chemotherapy (C1) (sex, age, anticipation of CINV, nausea terrain, history of nausea/vomiting, history of chemotherapy, motion sickness, tolerance of EO odour).
Compare and describe the use of antiemetics use of antiemetics | 1 month, 2 months and 3 months
  Compare and describe the use of antiemetics use of antiemetics and write down the use of EO inhalations EO inhalations "if needed" during the acute (D1), delayed (D4) and anticipated phase of CINV (H0) during the 3 cycles of chemotherapy (C1, C2 and C3).
Impact of inhaled aromatherapy on quality of life | 1 month, 2 months and 3 months
  Compare quality of life between the two groups at each each cycle of chemotherapy (C1,C2 and C3). Difference of quality of life score (EORTC QLQC30) between groups at each cycle.
  EORTC QLQC 30 is European Organisation for Research and Treatment of Cancer Quality of Life Core Questionnaire.
  This self-questionnaire, validated in French, assesses quality of life specific to cancer. It is intended for all cancer patients, regardless of location.
  EORTC QLQC 30 contains 30 items and assesses 15 dimensions of quality of life :
  * 5 functional scales: physical, cognitive, social, emotional or psychological and limitations in daily activities;
  * 1 global health/quality of life scale;
  * 9 symptom scales: tiredness, nausea and vomiting, pain, dyspnea, insomnia, loss of appetite, constipation and diarrhea, financial problems related with the disease.
Efficacy of inhaled aromatherapy on dietary intake | 1 month, 2 months and 3 months
  To compare the effect of inhalation of ginger + lemon EO versus placebo in addition to conventional antiemetic treatments on diet during C1, C2, C3. Difference of dietary intake measured by SEFI scale between groups.
  SEFI (Score d'Evaluation Facile des Ingesta - Ingesta Easy Evaluation Score) / LA description : SEFI is a visual assessment, by the patient himself or with the help of a caregiver, of his food intake, using an analog scale (0 to 10), or a choice of portions consumed.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CH BRIVE, Brivé
  - Chu La Reunion, La Réunion
  - University Hospital, Limoges, Limoges
  - Ch Poissy, Saint-Germain-en-Laye

IPD SHARING:
Plan to Share IPD: No